CLINICAL TRIAL: NCT02685436
Title: Role of Bronchoalveolar Lavage Pepsin Assay in Wheezy Infants
Brief Title: Role of Pepsin Assay in Wheezy Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Zaki, Lecturer, Mansoura University Children Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1722011
Record Dates: First submitted 2016-02-03; First posted 2016-02-18 (Estimated); Results first posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-09

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Omeprazole; Domperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- omeprazole and domperidone (Other): wheezy infants with GERD will receive 12 weeks of domperidone (0.2mg/kg/day t.d.s.) and omeprazole (10 mg/once/day).
  Interventions: Drug: Omeprazole and domperidone

INTERVENTIONS:
Drug: Omeprazole and domperidone — wheezy infants with abnormal MII-pH or reflux esophagitis will be given omeprazol(10mg/once/day) and domperidone (0.2mg/kg/day t.d.s)
  Other Names: omipak , motilium

SUMMARY:
Wheezy infants were tested for gastro-esophageal reflux disease (GERD) using combined multiple channel intraluminal impedance-pH (MII-pH), esophagogastroduodenoscope (EGD), lipid laden macrophage index and BAL pepsin. Wheezy infants with abnormal MII-pH or reflux esophagitis were given domperidone and omeprazole then re-evaluated for symptoms control and exacerbations recurrence.

DETAILED DESCRIPTION:
Wheezy infants were tested for gastro-esophageal reflux disease using combined MII-pH, EGD, LLMI and BAL pepsin. Wheezy infants with abnormal MII-pH or reflux esophagitis were given domperidone and omeprazole for 12 weeks then re-evaluated for symptoms control and wheeze exacerbations recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Infants with physician documented 3 attacks of wheezing episodes over the last 6 months or persistent wheeze over the last one month

Exclusion Criteria:

* Wheezy infants with atopy (allergic rhino-conjunctivitis or eczema), prematurity (less than 34 weeks), abnormal neurological examination, congenital heart diseases, airspace opacity on chest radiography, tracheal-bronchial malformations, immune deficiency and anatomical esophageal or gastric malformations

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2013-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tarek El-Desoky, Study Director — Faculty if medicine, Mansoura University

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: infants referred to the pediatric pulmonology unit at MUCH for evaluation because of recurrent or persistent wheeze were evaluated for the presence of GERD at gastro-enterology and hepatology unit.
Period: Overall Study
Arm/Group | Omeprazole and Domperidone
Started | 52 (the overall studied group)
Completed | 38 (GERD positive patients by either combined MII-pH or esophageal biopsy)
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | Omeprazole and Domperidone
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 52
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: months] | 9 [3 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 35
type of wheezing; persistent wheeze,intermittent wheeze [Count of Participants; unit: Participants] — persistent wheeze: wheeze for 1 month intermittent wheeze,: 3 wheeze episodes in 6 months
  Participants
    persistent wheeze | 27
    intermittent wheeze | 25
combined multiple channels intraluminal impedence-pH (MII-pH) monitoring [Count of Participants; unit: Participants] — positive combined multiple channels intraluminal impedence-pH (MII-pH) monitoring.
  negative combined multiple channels intraluminal impedence-pH (MII-pH) monitoring.
  Participants
    combined MII-pH positive | 34
    combined MII-pH negative | 18
esophageal biopsy [Count of Participants; unit: Participants] — reflux esophagitis no reflux esophagitis
  Participants
    reflux esophagitis | 18
    no reflux esophagitis | 34
Any positive test (combined MII-pH monitoring and/or endoscopic esophageal biopsy) [Count of Participants; unit: Participants] — positive combined MII-pH monitoring and/or endoscopic esophageal biopsy. negative combined MII-pH monitoring and/or endoscopic esophageal biopsy
  Participants
    positive | 38
    negative | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Each Level of Wheeze Control
Description: Number of Participants with controlled Wheezing Number of Participants with partially controlled Wheezing Number of Participants with uncontrolled wheezing
Time Frame: 3 months
Population: Abnormal esophageal impedance-pH and or reflux esophagitis
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Group: a wheezy infant with positive combined MII-pH and/or reflux esophagitis
Arm/Group | Treatment Group
Number analyzed (Participants) | 38
Participants
  controlled | 18
  partially controlled | 11
  non controlled | 9

ADVERSE EVENTS:
Time Frame: not collected
Description: "Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Omeprazole and Domperidone
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Non randomization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes